CLINICAL TRIAL: NCT05113888
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial of Qizhi Weitong Granules in the Treatment of Abdominal Pain Symptoms in Diarrhea-type Irritable Bowel Syndrome
Brief Title: Exploratory Study on Dosage of Qizhi Weitong Granules in the Treatment of Irritable Bowel Syndrome （IBS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR999-QZWT-IBS-01
Record Dates: First submitted 2021-10-20; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Qizhi Weitong granules; Irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The study was divided into three groups: Qizhi Weitong granule high-dose group, Qizhi Weitong granule low-dose group and placebo group
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qizhi Weitong granules high-dose group (Experimental): interventions：Qizhi Weitong granules Specification: 5.0g/bag，the drug content is equivalent to 2 bags of Qizhi Weitong granules (2.5g/ bag commercially available).
  Interventions: Drug: Qizhi weitong granules(High）
- Qizhi Weitong granules low-dose group (Experimental): interventions：Qizhi Weitong granules Specification: 5.0g/bag，the drug content is equivalent to 1 bag of Qizhi Weitong granules (2.5g/ bag commercially available).
  Interventions: Drug: Qizhi weitong granules(Low）
- The control group (Placebo Comparator): interventions：Qizhi Weitong granules placebo Specification: 5.0g/bag，Does not contain effective crude drug ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qizhi weitong granules(High） — take orally before meals, 1 bag each time, 3 times a day.
  Arms: Qizhi Weitong granules high-dose group
Drug: Qizhi weitong granules(Low） — take orally before meals, 1 bag each time, 3 times a day.
  Arms: Qizhi Weitong granules low-dose group
Drug: Placebo — take orally before meals, 1 bag each time, 3 times a day.
  Arms: The control group

SUMMARY:
The purpose of this study are as follows: 1) To evaluate the efficacy and safety of Qizhi Weitong granules in the treatment of diarrhea-type irritable bowel syndrome (IBS-D);2) To explore the dosage of Qizhi Weitong Granulesin treatment of IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnostic criteria of WESTERN medicine IBS-D;
* Aged 18-65 (including 18 and 65 years old) years;
* The mean weekly NRS score for abdominal pain (the most severe in the past 24 hours) was between 3.0 and 7.0 within the last week, and there were at least 2 days per week when fecal traits were classified as type 6 or 7;
* Informed consent, voluntary test.

Exclusion Criteria:

* Stool number of type 7 according to Bristol Stool Chart, more than 3 times per day;
* TCM syndrome was diagnosed as deficiency of spleen and kidney Yang syndrome；
* Patients who took emergency medication (Piveronium bromide tablets) more than the standard during admission period (more than 2 days per week on average)；
* Patients who have been diagnosed with organic diseases of digestive system, such as inflammatory bowel disease, intestinal tuberculosis, intestinal tumor, etc., or are still complicated with peptic ulcer and infectious diarrhea；
* Patients with similar symptoms of IBS, such as eosinophilic enteritis, collagenous enteritis, lactose intolerance, etc.
* Patients with intestinal diseases of digestive system, such as tuberculous peritonitis, cirrhosis, chronic pancreatitis, etc.
* Patients with systemic diseases affecting digestive tract function, such as hyperthyroidism or hypothyroidism, endometriosis, chronic renal insufficiency, autoimmune diseases, diabetes, etc.
* Previous gastrointestinal surgery (except for appendicitis);
* Patients with serious cardiovascular diseases, serious liver and kidney diseases, hematopoietic system diseases, tumor, neurological or psychiatric system diseases;
* Major anxiety (SAS score ≥70) or major depression (SDS Score ≥73);
* Concomitant drugs affecting gastrointestinal motility and function (prokinetic drugs, anticholinergic drugs, calcium channel blockers, 5-HT3 receptor antagonists, antidiarrhea agents, antacids, antidepressants, antianxiety drugs, intestinal microbiota regulators, antibiotics, etc.) should not be discontinued in the test;
* Pregnant or lactating women who had a birth plan from enrollment to 3 months after the end of the trial.
* Allergic to the test drug emergency drug and its ingredients;
* Suspected or confirmed history of alcohol or drug abuse;
* Patients who participated in other clinical trials within 1 month prior to enrollment;
* Other subjects considered unsuitable for clinical trials by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain intensity | Recorded daily by patients from baseline to day56
  the most severe abdominal pain score in the past 24 hours, with a weekly mean decrease of at least 30% from baseline;
Improvement of stool characteristics | Recorded daily by patients from baseline to day56
  Record daily by symptom diary card.Stools were recorded according to Bristol Stool Chart.

SECONDARY OUTCOMES:
Frequency of abdominal pain | Recorded daily by patients from baseline to day56
  Number of abdominal pain
IBS symptom severity scale（IBS-SSS） | Baseline and days 14，28，56
  The IBS symptom severity questionnaire consists of four questions on a 100-point scale, with the highest score being 100 and the lowest being 0. The higher the score, the more severe the symptoms.
IBS Quality of Life Scale（IBS-QOL） | Baseline and days 14，28，56
  The IBS Quality of Life scale has 34 questions, and adopts a five-level scoring system, with the highest score of 4 points and the lowest score of 0 points. The higher the score, the more serious it is.
Self-rating Anxiety Scale（SAS) | baseline and day56
  There are 20 questions in the self-rating anxiety scale, which is graded at four levels, with the highest score being 4 and the lowest score being 1. The higher the score is, the more serious it is.
Self-rating Depression Scale(SDS) | baseline and day56
  There are 20 questions in the Self-rating Depression Scale, which is graded at four levels, with the highest score being 4 and the lowest score being 1. The higher the score is, the more serious it is.
Emergency drug use | Emergence，baseline and days 14，28，56
  Subjects may take Piaverium bromide tablets 3-4 tablets per day if they feel unbearable abdominal pain, and increase to 6 tablets per day if necessary.

IPD SHARING:
Plan to Share IPD: No